CLINICAL TRIAL: NCT07067476
Title: A Randomized, Double-Blind, Split-Face Clinical Study to Evaluate the Redness Relief Efficacy of Instant Flush Products in Subjects With Sensitive Skin
Brief Title: Instant Flush Redness Clinical Efficacy Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C25005021
Record Dates: First submitted 2025-07-03; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Sensitive Skin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Side: Instant Anti-Redness Emulsion (Experimental): Participants will receive 0.3g of test emulsion (FLA#2039188 43) applied to one half of their face. The emulsion contains panthenol (Vitamin B5 precursor) and is designed to reduce facial redness after infrared heat-induced stimulation.
  Interventions: Other: Instant Anti-Redness Emulsion (FLA#2039188 43)
- Control Side: Water Only (Placebo Comparator): Participants will receive 0.3g of purified water applied to the opposite side of the face, serving as control. Redness relief will be compared between the test emulsion and water using clinical assessment and imaging tools.
  Interventions: Other: Purified Water (Control)

INTERVENTIONS:
Other: Instant Anti-Redness Emulsion (FLA#2039188 43) — A topical emulsion not yet marketed, developed to relieve skin redness. It contains panthenol and is applied once to the test side of the face after heat-induced redness.
  Arms: Test Side: Instant Anti-Redness Emulsion
Other: Purified Water (Control) — 0.3g of water is applied to the control side of the face. Used as placebo comparator to evaluate the redness-relieving efficacy of the test emulsion.
  Arms: Control Side: Water Only

SUMMARY:
The goal of this clinical trial is to learn if an anti-redness emulsion can help lower facial redness caused by heat in healthy adult women. The main questions it aims to answer are:

* Does the anti-redness emulsion lower facial redness better than purified water?
* Is the product safe and comfortable to use?

Researchers will compare the anti-redness emulsion to purified water using a split-face method.

Participants will:

* Receive infrared light on their face to trigger redness
* Apply the anti-redness emulsion to one side of their face and purified water to the other side
* Have their facial redness measured at different time points using photography, imaging devices, and skin redness tests
* Answer questions about their experience with the products

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged from 20-40 years old.
2. Self-declared mild sensitive skin.
3. Self-declare with skin concerns of redness and easy to flush.
4. Willing to be exposed to infrared light on the facial skin to induce facial redness(can tolerate heat sensation on the face).
5. Clinical grading of skin redness (visual) ≥ 4 after infrared light induction (7-8 mins) by dermatologist.
6. No disagreement of dermatologist because of other reasons that exclude the parficipation of the subject.
7. In general good health at the time of the study.
8. Willing and able to participate as evidenced by signing of informed consent and photo release

Exclusion Criteria:

1. Allergic to infrared light
2. Pregnant or breast-feeding woman or woman planning pregnancy during the study.
3. Subject deprived of rights by a court or administrative order.
4. Major subject to a guardianship order.
5. Subject residing in a health or social care establishment.
6. Patient in an emergency setting
7. Subject with a skin disease in the test areas (particularly e.g, acne, rosacea, eczema).
8. Subjects with history, of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, medication, cosmetic: or personal care products or ingredients.
9. Subject presenting a stable or progressive serious disease (per investigator's assessment).
10. Immuno-compromised subject.
11. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
12. Subjects regularly practicing aquatic or nautical sports.
13. Subjects regularly attending a sauna.
14. Subject with cardiovascular or circulatory history.
15. Subject with a history of skin cancer or malignant melanoma.
16. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in skin redness visual score (Griffith 10-point scale) | Baseline to 2 hours post-application
  Skin redness will be assessed by a dermatologist using the Griffith visual 10-point scale on the left and right sides of the face. Higher scores on the Griffith 10-point scale indicate greater skin redness, which is considered a worse outcome. Assessments will occur at Tbefore (before infrared induction), T0 (after infrared induction), T10min (10 mins post-application), T1h (1 hour post-application), and T2h (2 hours post-application).

SECONDARY OUTCOMES:
Change in facial redness area ratio (Visia 7 image analysis) | Baseline to 2 hours post-application
  Standard and polarized images of the face will be captured by Visia 7. The red area ratio will be calculated from red mode images before and after product application.
Change in erythema index (Mexameter® MX 18) | Baseline to 2 hours post-application
  Erythema index will be measured based on spectral absorption at both sides of the cheeks. Measurements will be taken at Tbefore, T0, T10min, T1h, and T2h.
Change in red blood cell (RBC) concentration measured by TiVi 700 | Baseline to 2 hours post-application
  The TiVi 700 Tissue Viability Imaging System will be used to assess RBC concentration in the facial skin as a marker of microcirculation. Measurements will be taken before and after infrared induction and at multiple timepoints after product application.
Change in facial skin temperature measured by thermal imaging (Fluke TiS60+) | Baseline to 2 hours post-application
  Thermal images of both sides of the cheek will be captured by Fluke TiS60+ to evaluate skin temperature changes in response to product application. Images will be taken at multiple timepoints from before infrared induction to 2 hours post-application.
Subject self-assessment of product efficacy and tolerance | 15 minutes post-application
  Participants will complete self-assessment questionnaires 15 minutes after product application to evaluate perceived product efficacy and tolerance, including redness reduction and skin comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon study completion and PRS registration completion.
  Timeline:
  Months 2-3: Data de-identification, metadata preparation, and platform integration.
  Month 4: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn